CLINICAL TRIAL: NCT04968860
Title: Clinical-microbiological Study of Oral Health Condition and Quality of Life of Children/Adolescent With Acute Lymphoid Leukemia and Acute Myeloid
Brief Title: Oral Health Condition and Quality of Life in Children With Leukemia
Status: Terminated | Type: Observational
Why Stopped: Low casuistry that did not allow the study to continue
Sponsor: Paulo Sergio da Silva Santos (Other)
Responsible Party: Sponsor-Investigator, Paulo Sergio da Silva Santos, Associate Professor of the Department of Surgery, Stomatology, Pathology and Radiology - Bauru School of Dentistry - University of São Paulo, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Other Study IDs: LEUKEMIARAQ
Record Dates: First submitted 2020-06-03; First posted 2021-07-20 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Leukemia, Lymphoblastic; Leukemia, Myeloid, Acute
Keywords: Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Microbiota; Mouth; Quality of life; Children
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — There are going to collect saliva for this study, which is going to be stored for 10 years as the maximum limit.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Composed of children/adolescent individuals who have a definitive diagnosis of lymphoid leukemia or acute myeloid leukemia, who will be invited to participate in the research, regardless of race or gender.
  Interventions: Other: This study is observational
- Control group: The control group is going to consist of healthy children/adolescent individuals, non-syndromic, without history of cancer, matched by age and gender in relation to the study group, who have not used antibiotics 48 hours before or in the day of evaluation.
  Interventions: Other: This study is observational

INTERVENTIONS:
Other: This study is observational — * Clinical evaluation of the oral health condition
  * Microbiota evaluation by analyzing the collected saliva
  * Application of questionnaires of quality of life

SUMMARY:
Among the different types of cancer that most affect children, leukemia is the principal. One of the main treatments for leukemia is chemotherapy. Among the most common side effects of chemotherapy are nausea and/or vomiting, diarrhea, fatigue, alopecia, neuropathy, opportunistic infections, and oral mucositis. It is still necessary to establish which microorganisms are predominant in the oral microbiota of children with leukemia, which factors influence it, what is its relationship with oral mucositis and what is their impact in the quality of life. To better understand the risks of secondary infection, it is important to develop preventive and/or therapeutic strategies to control the side effects of antineoplastic treatment in the mouth that may negatively impact the quality of life, to expose the risk of death as well as raise hospital costs for the care of children with leukemia. Objective: To identify the clinical characteristics of the oral condition, types of microorganisms of the oral microbiota, and quality of life in children/adolescents with acute lymphoid leukemia and acute myeloid leukemia before and during antineoplastic treatment, and compare them with healthy children/adolescent individuals. Methodology: Longitudinal, case-control study, with a convenience sample. The study group, composed of children/adolescent individuals who have a definitive diagnosis of acute lymphoid leukemia or acute myeloid leukemia. The control group, non-syndromic children/adolescents, with no history of cancer, matched by age and gender. The clinical condition of the mouth will be evaluated by means of indexes: dental caries index (dmft index), gingival index (GA), and simplified oral hygiene index. The assessment of the quality of life through the ohip-14 and POS-version14 quality of life questionnaire and microbiological evaluation of saliva through MALDI-TOF analysis. Statistical analysis will be performed through relative risk for cohort study with more than three paired groups. Odds ratio, for the control group more than three controlled groups and Mcnemere, for comparison with the control group, for more than three paired groups.

DETAILED DESCRIPTION:
In children, non-communicable diseases such as cancer are increasing every year. It became a priority on the global child health agenda. Each year, there were an estimated 30.000 new cases of cancer in children/adolescent individuals. In Brazil, between 2018-2019, there were 12.500 new cases of cancer in children and adolescents up to 19 years of age. The mortality rate was 7.917 cases.

Among the types of cancer that most affect children, leukemia is the most prevalent. In 2018, there was a forecast of 437.033 new cases of leukemia with a mortality of 309.006 individuals around the world.

One of the main treatments for leukemia is chemotherapy, the side effects can affect different parts of the body that may present since the beginning of the treatment. Chemotherapy produces systemic toxicity resulting in anemia, leukopenia, and thrombocytopenia that is more intense in the treatment of oncohematological diseases when compared to solid tumors. Among the most common side effects of chemotherapy are included nausea and/or vomiting, diarrhea, fatigue, alopecia, neuropathy, opportunistic infections, and oral mucositis.

Some studies reported that the intensity of oral mucositis, as well as the risk of sepsis from secondary infection in the mouth of individuals with cancer, they can be influenced by some specific microorganisms present in the oral cavity. Factors such as oral hygiene, presence of dental caries, and periodontal disease may be related to the type of microorganisms present in the oral cavity. There is a lack of studies about microbiota oral in leukemic children. Oral microbiota in children with leukemia is predominantly composed of gram-positive microorganisms such as Streptococus viridans, Streptococous mutans and Lactobacillus when compared to adults oral microbiota where gram-negatives microorganisms such as Klebsiella spp., E coli, Enterobacter, Pseudomonas spp. predominate. It is noteworthy that it is necessary to establish what kind of microorganisms are predominant in the oral microbiota of children with leukemia, also which factors influence it, and what is the relationship among the oral mucositis, general clinical status, and quality of life of the children/adolescent with cancer.

Therefore, it is important to identify the risks of secondary infection in oral cavity, to be able to develop preventive and/or therapeutic strategies to control the side effects of antineoplastic treatment in the mouth that can negatively impact the quality of life, expose the risk of death as well as raise hospital costs for the care of children with leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who, based on the agreement of parents and/or guardians, agree to participate in the research with a signed "Informed Consent Form"
* Patients from 3 to 17 years of age
* Patients older than 6 years must not only have parental and/or guardian authorization must have the consent term
* Patients who have not started antineoplastic treatment
* Patients with ALL only with BFM protocol
* AML patients with BFM protocol only

Exclusion Criteria:

* Responsible for patients who do not sign the free and informed consent form.
* Patients under three years of age and over 17 years of age
* Children older than six years who do not agree to the term of assent
* Patients who have started antineoplastic treatment
* Patients with syndromes and/or other systemic diseases associated with the diagnosis of lymphoid and acute myeloid leukemia
* Neoplasms other than lymphoid leukemia or acute myeloid

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study group will be composed of children/adolescent individuals who have a definitive diagnosis of lymphoid leukemia or acute myeloid leukemia, who will be invited to participate in the research, regardless of race or gender.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2022-12-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of dental condition | 5 minutes to 10 minutes
  Dental condition is going to be evaluated by dental caries index (dmft index) (WHO, 2013).
Evalulation of periodontal condition | 10 minutes to 15 minutes
  The periodontal evaluation it is goning to be evaluated by and gingival index (LOE, 1964)
Evalulation of oral hygiene | 10 minutes to 15 minutes
  Oral hygiene is going to be evaluated by simplified oral hygiene index (IHO-S).
To evaluate oral mucositis | 5 minutes to 10 minutes
  the presence of oral mucositis will be evaluated through the graduation recommended by the World Health Organization (WHO) (WHO, 1979).
Evaluation of oral pain of oral mucositis | 1 minutes to 2 minutes
  The oral pain because of the oral mucositis is going to be evaluated by Visual Analogue Scael of pain and it is gonig to be scaled by the Wong-Backer face scale which is from 0 to 10 pontuation, being 1 the minimium pain percivied and 10 de maximium pain percieved. This evaluation it is going to be make only in children with leukemia.
Saliva collection | 15 minutes to 20 minutes
  The collection of the saliva is going to be made by an unstimulated technic. The minimum of 2 mL to maximum of 10 ml of saliva are going to be collected.
to evaluate the quality of life of children percieved by parents | 10 to 15 minutes
  A Pediatric Quality of Life Inventory Version 4.0 questionaire is going to be answered by children parentes with the following five options: never = 0, almost never = 1, sometimes = 2, often = 3, and almost always = 4.
to evaluate the impact of oral condition on the quality of life percieved by the children | 10 to 15 minutes
  A OHIP-14 (Oral Health Impact Profile) questionnaire (adapted for children) is going to be applied to children with 6 years old or children older than 6 years old. The questionaire is going to be answered with five options: never = 0, almost never =1 , sometimes = 2, often = 3, and almost always = 4 which is represented by a face scale.

CONTACTS AND LOCATIONS:
Overall Officials: Reyna A Quispe, MsC, Principal Investigator — Faculdade de Odontologia de Bauru, Universidade de São Paulo
Locations (1):
- Faculdade de Odontologia de Bauru, Universidade de São Paulo, Bauru, São Paulo, Brazil

REFERENCES:
- [Background] Steliarova-Foucher E, Fidler MM, Colombet M, Lacour B, Kaatsch P, Pineros M, Soerjomataram I, Bray F, Coebergh JW, Peris-Bonet R, Stiller CA; ACCIS contributors. Changing geographical patterns and trends in cancer incidence in children and adolescents in Europe, 1991-2010 (Automated Childhood Cancer Information System): a population-based study. Lancet Oncol. 2018 Sep;19(9):1159-1169. doi: 10.1016/S1470-2045(18)30423-6. Epub 2018 Aug 8. PMID 30098952
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Carlotto A, Hogsett VL, Maiorini EM, Razulis JG, Sonis ST. The economic burden of toxicities associated with cancer treatment: review of the literature and analysis of nausea and vomiting, diarrhoea, oral mucositis and fatigue. Pharmacoeconomics. 2013 Sep;31(9):753-66. doi: 10.1007/s40273-013-0081-2. PMID 23963867
- [Background] Ozdemir ZC, Bozkurt Turhan A, Duzenli Kar Y, Dinleyici CE, Bor O. Fatal course of Saprochaete capitata fungemia in children with acute lymphoblastic leukemia. Pediatr Hematol Oncol. 2017 Mar;34(2):66-72. doi: 10.1080/08880018.2017.1316808. Epub 2017 Jun 2. PMID 28574735
- [Background] Damascena LCL, de Lucena NNN, Ribeiro ILA, de Araujo TLP, de Castro RD, Bonan PRF, Lima Neto EA, de Araujo Filho LM, Valenca AMG. Factors Contributing to the Duration of Chemotherapy-Induced Severe Oral Mucositis in Oncopediatric Patients. Int J Environ Res Public Health. 2018 Jun 1;15(6):1153. doi: 10.3390/ijerph15061153. PMID 29865201
- [Background] Napenas JJ, Brennan MT, Bahrani-Mougeot FK, Fox PC, Lockhart PB. Relationship between mucositis and changes in oral microflora during cancer chemotherapy. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Jan;103(1):48-59. doi: 10.1016/j.tripleo.2005.12.016. Epub 2006 Apr 21. PMID 17178494
- [Background] Santos de Faria AB, Silva IH, de Godoy Almeida R, Silva SP, Carvalho AT, Leao JC. Seroprevalence of herpes virus associated with the presence and severity of oral mucositis in children diagnosed with acute lymphoid leukemia. J Oral Pathol Med. 2014 Apr;43(4):298-303. doi: 10.1111/jop.12138. Epub 2013 Dec 10. PMID 24325331
- [Background] O'Sullivan EA, Duggal MS, Bailey CC, Curzon ME, Hart P. Changes in the oral microflora during cytotoxic chemotherapy in children being treated for acute leukemia. Oral Surg Oral Med Oral Pathol. 1993 Aug;76(2):161-8. doi: 10.1016/0030-4220(93)90198-d. PMID 8361725
- [Background] Volpato LE, Kloster AP, Nunes LF, Pedro FL, Borges AH. Cariogenic microbiota of children under chemotherapy: A pilot study. J Indian Soc Pedod Prev Dent. 2016 Oct-Dec;34(4):370-6. doi: 10.4103/0970-4388.191423. PMID 27681402
- [Background] Valera MC, Noirrit-Esclassan E, Pasquet M, Vaysse F. Oral complications and dental care in children with acute lymphoblastic leukaemia. J Oral Pathol Med. 2015 Aug;44(7):483-9. doi: 10.1111/jop.12266. Epub 2014 Sep 22. PMID 25243950
- [Background] Wang Y, Xue J, Zhou X, You M, Du Q, Yang X, He J, Zou J, Cheng L, Li M, Li Y, Zhu Y, Li J, Shi W, Xu X. Oral microbiota distinguishes acute lymphoblastic leukemia pediatric hosts from healthy populations. PLoS One. 2014 Jul 15;9(7):e102116. doi: 10.1371/journal.pone.0102116. eCollection 2014. PMID 25025462
- [Background] Villafuerte KRV, Martinez CJH, Dantas FT, Carrara HHA, Dos Reis FJC, Palioto DB. The impact of chemotherapeutic treatment on the oral microbiota of patients with cancer: a systematic review. Oral Surg Oral Med Oral Pathol Oral Radiol. 2018 Jun;125(6):552-566. doi: 10.1016/j.oooo.2018.02.008. Epub 2018 Feb 21. PMID 29566996
- [Background] Bardellini E, Amadori F, Majorana A. Oral hygiene grade and quality of life in children with chemotherapy-related oral mucositis: a randomized study on the impact of a fluoride toothpaste with salivary enzymes, essential oils, proteins and colostrum extract versus a fluoride toothpaste without menthol. Int J Dent Hyg. 2016 Nov;14(4):314-319. doi: 10.1111/idh.12226. Epub 2016 May 10. PMID 27160933
- [Background] Grando LJ, Mello ALSF, Salvato L, Brancher AP, Del Moral JAG, Steffenello-Durigon G. Impact of leukemia and lymphoma chemotherapy on oral cavity and quality of life. Spec Care Dentist. 2015 Sep;35(5):236-242. doi: 10.1111/scd.12113. Epub 2015 May 12. PMID 25963973